CLINICAL TRIAL: NCT05848973
Title: The NutriMind Trial: A Low-cost Randomized Trial Combining a Healthy Diet and Psychotherapy to Treat Depressive Symptoms Among University Students - The Case of Uganda
Brief Title: NutriMind: A Combination of Healthy Diet and Psychotherapy to Treat Depression
Acronym: NutriMind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: University of Oslo (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Prudence Atukunda Friberg, Associate Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 441814
Record Dates: First submitted 2023-03-27; First posted 2023-05-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Diet, Healthy; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: The NutriMind trial will include three intervention groups, namely; the healthy diet group, the psychotherpay group (Mindfulness-Based Cognitive Therapy-MBCT), a combined healthy diet and MBCT group and a control group with no intervention. Pending the financial situation investigators may also consider having two arms: Intervention (Diet and MBCT) and control.
Who Masked: Outcomes Assessor
Masking Description: The data collection teams will be blinded to the allocation arms throughout the trial in order to minimise measurement bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy diet (Active Comparator): The study participants randomized to this arm will be given advice about consuming a healthy diet, i.e. a diet rich in vegetables/fruits and wholegrain/fibre, fish, olive oil; and moderate in red meat and dairy products. The participants will receive 8 weekly, one hour group sessions delivered by trained nutritionists.
  Interventions: Other: Healthy Diet
- Mindfulness-based cognitive therapy (MBCT) (Active Comparator): The study participants randomized to this arm will be taught the purpose and application of MBCT, namely to modify cognitive and effective processes in the management of depressive symptoms as well as relapse prevention among those with residual depressive symptoms. It is a structured 8-weeks' intervention program delivered in groups, with an all-day practice session around week six and regular reunion sessions thereafter.
  Interventions: Behavioral: Mindfulness-based cognitive therapy (MBCT)
- Healthy diet and MBCT combined (Active Comparator): The study participants randomized to this arm will receive both the healthy diet intervention and the MBCT intervention
  Interventions: Other: Healthy Diet; Behavioral: Mindfulness-based cognitive therapy (MBCT)
- Control (No Intervention): No particular intervention will be provided to the control group.

INTERVENTIONS:
Other: Healthy Diet — The targeted study participants will be given advice about healthy dietary intakes. This will entail promotion of foods rich in vegetables/fruits and wholegrain/fibre, fish, olive oil; moderate in lean red meat and low-fat diary products). To be concrete, the study investigators will target energy (E%) from macronutrients as follows: 42 E% total fat (≥ 22 E% from monounsaturated fatty acids, 10 E% from polyunsaturated fatty acids and <10 E% saturated fatty acids), 35 E% carbohydrate, 15 E% protein and ≤ E 5% alcohol. Importantly, this will meet all Recommended Dietary Intake requirements for adults.
  Arms: Healthy diet; Healthy diet and MBCT combined
Behavioral: Mindfulness-based cognitive therapy (MBCT) — MBCT is a skills-based intervention comprising a structured 8-week group intervention program to be delivered in groups of study participants, with an all-day practice session around week six and regular reunion sessions thereafter.
  Arms: Healthy diet and MBCT combined; Mindfulness-based cognitive therapy (MBCT)

SUMMARY:
University students in Low- and Middle-Income Countries (LMIC) continue to face growing rates of depression, a common mental health problem. Adding to this burden is the mental health treatment gap, necessitating the need to identify new treatment methods that can easily be implemented at a large scale.

This project will test if a healthy diet combined with mindfulness-based cognitive therapy can reduce depressive symptoms among university students in Uganda, a low resource country.

The burden of depression is high in sub-Saharan African countries, largely worsened by poverty, hunger and poor public health service, and lately the COVID-19 pandemic. These factors increase psychological distress among young people in sensitive periods of life, such as students who are about to choose their career and establish family. Successfully managing depression in LMIC is likely to depend on low-cost treatment that can easily be managed to large target populations, yet still be at the scientific forefront, proof-based, and culturally acceptable. This can possibly be obtained with an intervention combining healthy diet and cognitive behavioral therapy based on mindfulness principles.

While healthy diets and mindfulness cognitive therapy individually can partly lessen the burden of depression, these two therapeutic modalities have not been tested in combination among university students in sub-Saharan Africa, i.e. a synergistic effect that is still to be studied.

With the NutriMind Trial, its investigators focus on a neglected global mental health challenge, namely depression among university students in Uganda.

DETAILED DESCRIPTION:
Despite being a major global health issue for decades, Common Mental Health Problems (CMHPs), such as depression, remains neglected. University students worldwide are facing growing rates of CMHPs, with few or no mental health services available. The burden of CMHPs is highest in low- and middle-income countries (LMICs), largely worsened by poverty, hunger and poor public health governance. These factors increase stress, in particular among students who are about to choose their career, both in academia and later in the work force. Successfully managing CMHPs in LMICs is likely to depend on treatment methods that can easily be administered to the target population, yet still be at the scientific forefront, evidence-based, and culturally acceptable.

Wellness-based therapy includes behavioural changes like mindfulness-based cognitive therapies and nutritional interventions. While systematic reviews and randomized controlled trials show that such treatment modalities may lessen the burden of CMPHs, including depression, they have not been tested among university students in LMICs. The NutriMind investigators will therefore perform a randomized controlled trial to test if mindfulness-based cognitive therapy and/or a healthy diet (modified Mediterranean diet) will reduce depressive symptoms among university students in Uganda, a low-income country. In addition to evaluate the clinical outcomes, the investigators will analyse biomarkers for various metabolic pathways, as studies have related e.g. inflammation and oxidative stress to depression. Recent studies also indicate that the microbiome can play a role in depression through orchestrating metabolic signals to the brain. Notwithstanding these ambitious goals, our experienced and cross-disciplinary team puts us in an advantageous position to successfully accomplish this work.

The overall goal of the project is thus to test pragmatic lifestyle interventions in a population at high risk of depression in a low-resource setting and link the study outcomes to biological processes. If the investigators succeed, they can readily identify those who will improve from the intervention and provide an opportunity to respond to current gaps in mental health treatment, in particular in LMICs. In doing so, this novel project will address the World Health Organization's appeal for immediate and sustained action to reduce mental health illnesses, and the Lancet Commission's call for a substantial global shift toward healthy dietary patterns, as well as United Nations Sustainable Development Goals, in particular nos. 3 (good health and well-being) and 4 (quality education).

ELIGIBILITY:
Inclusion criteria:

* Those who score between 16 and 25 on the CES-D scale
* Completed >1 study-year of study and have >2 study-years before graduation
* Not using any medication regularly that might interfere with study adherence or - outcomes
* Giving consent to participate

Exclusion criteria:

* Not being diagnosed with chronic disorder or cancer
* Not being pregnant
* Not having food allergy- or intolerance
* Not having experienced recent bereavement or major personal loss (e.g. income or divorce)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 24 months in depressive symptoms using the Center for Epidemiological Studies - Depression (CES-D) score among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Depressive symptoms will be assessed using the CES-D score from before to after the intervention. CES-D scores range from 0 to 60, with higher scores indicating greater depressive symptoms. The CES-D provides cut-off scores (16 or greater) to aid in identifying individuals at risk for clinical depression, with good sensitivity and specificity and high internal consistency.

SECONDARY OUTCOMES:
Change from baseline to 24 months in depressive symptoms using the Beck Depression Inventory-II (BDI-II) score among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  BDI-II is a self-reported, validated tool for screening depressive symptoms on a 4-point scale with 21 questions, giving a range of 0-63. A score > 10 strongly indicates depression.
The health economic costs of each of the three intervention arms compared with the control group. | 24 months
  Health economic costs of the interventions on change in depressive symptoms will be evaluated using standard cost-effectiveness methods including sensitivity analysis. Investigators will convert the CES-D and BDI-II scores into a generic health measure (e.g. disability/quality adjusted life years) for this purpose.
Change from baseline to 24 months in body weight among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Weight in kilograms will be measured using a scale (to the nearest 100 g)
Change from baseline to 24 months in body height among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Height in meters will be measured using a scale (to the nearest cm)
Change from baseline to 24 months in body composition among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Body composition (i.e. percentage of fat, bone, water and lean body mass) will be assessed with bio-impedance.
Change from baseline to 24 months in blood cholesterol levels among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Blood cholesterol (mmol/l) will be analyzed using standard biochemistry methods, levels above the reference range indicate increased risk of cardiovascular disease.
Change from baseline to 24 months in blood CRP levels among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Blood CRP (mg/l) will be analyzed using standard biochemistry methods, levels above the reference range indicate increased risk of cardiovascular disease.
Change from baseline to 24 months in fecal microbiota composition levels among the study participants randomized to each of the three intervention arms compared with the controls. | 24 months
  Microbiota (percentage distribution of various bacteria) will be analysed feces using 16S rRNA amplicon sequencing. Less diverse microbiota composition may indicate increased risk of depression and other non-communicable diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Prudence A Friberg, Principal Investigator — University of Bergen
Locations (1):
- Makerere University, Kampala, Central Uganda, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Informed Consent Form (ICF) will be shared with all study participants and was approved by Uganda Institutional Review Board.
  Clinical Study Report (CSR) will be published on the trial website that is going to be created during the study.
  There is signed Material Transfer Agreement (MTA) between the collaborating universities that specifies data sharing process
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Approximately 3 years from the start of the study.When all collected data has been analysed and published the results in an open access journal.
Access Criteria: Project website that will be established when the study implementation starts

REFERENCES:
- [Derived] Kardel KR, Iversen PO, Kaaya AN, Muhoozi G, Veierod MB, Wangen KR, Borosund E, Friberg PA. A pragmatic randomized trial to examine the effect of combining healthy diet with mindfulness cognitive therapy to reduce depressive symptoms among university students in a low-resource setting: protocol for the NutriMind Project. BMC Psychiatry. 2024 Sep 11;24(1):610. doi: 10.1186/s12888-024-06056-9. PMID 39261786